CLINICAL TRIAL: NCT00191230
Title: A Randomized Phase II Trial of Gemcitabine Containing Regimens (Gemcitabine/Carboplatin and Gemcitabine/ Cisplatin)When Used as Preoperative Chemotherapy for Patients With Stage I and II NSCLC
Brief Title: Gemcitabine/Platinum Containing Regimens as Preoperative Chemotherapy for Patients With Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5489; B9E-US-S236
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Cisplatin

INTERVENTIONS:
Drug: gemcitabine
Drug: carboplatin
Drug: cisplatin

SUMMARY:
To study the efficacy and tolerability of gemcitabine/platinum chemotherapy in non small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically of cytologically confirmed non small cell lung cancer
* No prior chemotherapy or radiation
* No prior malignancy

Exclusion Criteria:

* Pregnant or breastfeeding
* Serious concomitant systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2001-09; Study Completion 2006-07

PRIMARY OUTCOMES:
Complete pathological response

SECONDARY OUTCOMES:
Response rate, disease free survival, toxicity including pulmonary toxicity,operative mortality and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina, United States